CLINICAL TRIAL: NCT03503266
Title: An Open-label, Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C]-MT-7117 After a Single Oral Dose to Healthy Male Subjects
Brief Title: Mass Balance Study With MT-7117
Acronym: MT-7117 MB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MT-7117-E02; 2017-004549-25 (EudraCT Number)
Record Dates: First submitted 2018-03-18; First posted 2018-04-19 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteer
Keywords: Mass Balance Study with MT-7117

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] MT-7117 (Experimental): 14-C MT-7117
  Interventions: Drug: [14C] MT-7117

INTERVENTIONS:
Drug: [14C] MT-7117 — 14-C MT-7117

SUMMARY:
This is a single-centre, open-label, mass balance study in healthy male subjects utilising a single oral dose of [14C] MT 7117.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to provide written informed consent to participate in this study after reading the participant information sheet and Informed Consent Form, and after having the opportunity to discuss the study with the Investigator or designee.
* 2. Caucasian male subjects aged 30 to 65 years (inclusive) at Screening.
* 3. Healthy and free from illness or disease as determined by medical history, physical examination, electrocardiogram (ECG), vital signs, laboratory and other tests at Screening and Day -1, unless deemed not clinically significant by the Investigator or designee.
* 4. Body weight of 60 to 110 kg (inclusive) and a body mass index (Quetelet index) ranging from 18 to 32 kg/m2 (inclusive) at Screening and Day -1.
* 5. Vital signs within the following ranges at Screening and Day -1:

  * Systolic blood pressure: 90 to 140 mmHg
  * Diastolic blood pressure: 50 to 90 mmHg
* 6. Subjects and partners agree to use contraception throughout the study, as defined in the Protocol body.
* 7. Able to understand, in the Investigator's opinion, the nature of the study and any risks involved in participation and willing to cooperate and comply with the Protocol restrictions and requirements.
* 8. Regular daily bowel movements (i.e., production of at least one stool per day).

Exclusion Criteria:

* 1. Presence or history of severe adverse reaction or allergy to any medicinal product that is of clinical significance.
* 2. Participated in more than three clinical studies of a new chemical entity in the previous year or participated in a clinical study of any IMP within 12 weeks or five half-lives (whichever is longer) before the administration of IMP in this clinical study.
* 3. Consumption of any food-supplements, prescribed or over the counter medicine (including herbal and dietary supplements, such as St. John's Wort) during the 7 days (or 14 days if the medicine is a potential enzyme inducer) or five half-lives (whichever is longer) before the administration of IMP and during the study, unless in the opinion of the Sponsor and the Investigator, the medication will not interfere with the objectives of the study or compromise the subject's safety (Note: The use of acetaminophen [2 g/day for up to 3 consecutive days] will be permitted from Screening and during the study).
* 4. Clinically significant (in the opinion of the Investigator) endocrine, thyroid, hepatic (including Gilbert's syndrome), respiratory, gastrointestinal or renal disease, diabetes mellitus (type I and II), coronary heart disease, hypertension, or significant history of any psychiatric/psychotic disorder (including anxiety, depression and reactive depression).
* 5. Clinically relevant abnormal medical history, physical findings or laboratory values at Screening or Day -1 that could interfere with the objectives of the study or the safety of the subject, as judged by the Investigator.
* 6. Subjects with aspartate aminotransferase or alanine aminotransferase ≥2 x upper limit of normal or bilirubin above reference range at Screening or Day -1, confirmed by a repeat test at each visit.
* 7. Has a positive hepatitis B surface antigen, hepatitis B core antibody, hepatitis C virus antibody, or human immunodeficiency virus type 1 (HIV-1) and type 2 (HIV-2) result at Screening.
* 8. Clinically significant abnormal 12-lead ECG findings, including subjects with corrected QT interval using Fridericia's formula (QTcF) of >450 ms, or presence of atrial fibrillation or other significant arrhythmia at Screening or Day -1, confirmed by repeat assessment.
* 9. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardise the subject in case of participation in the study. The Investigator should be guided by evidence of any of the following:

  * history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding;
  * history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bowel resection;
  * history or clinical evidence of pancreatic injury or pancreatitis.
* 10. Excessive consumption of food or drink containing caffeine, including coffee, tea, cola, energy drinks or chocolates (>5 cups of coffee or equivalent per day).
* 11. Consumption of food or drink containing grapefruit, poppy seeds or Seville oranges from 7 days before the administration of the IMP.
* 12. Presence or history (in the last 2 years) of alcohol abuse or weekly alcohol intake of more than 28 units (224 g) or a positive urine or breath alcohol test at Screening or Day 1. One unit (8 g) is equivalent to a ½ pint (280 mL) of beer, 1 measure (25 mL) of spirits or 1 small glass (125 mL) of wine.
* 13. Presence or history of drug abuse (as defined by Diagnostic and Statistical Manual of Mental Disorders [DSM-V] criteria) or a positive urine test for drugs of abuse at Screening or Day -1.
* 14. Donation of one or more units of blood (450 mL) within 3 months before the administration of the IMP, or plasma within 7 days prior to Screening, or platelets within 6 weeks prior to Screening or the intention to donate blood within 3 months after the final study visit.
* 15. Use of tobacco or nicotine-containing products (snuff, chewing tobacco, cigars, pipes, e cigarettes or nicotine replacement products) within the 3 month period prior to administration of IMP, during the confinement period and until the final study visit, or positive urine cotinine test at Screening or Day -1.
* 16. Heavy physical training or excessive exercise (e.g., long distance running, weight lifting or any physical activity to which the subject is not accustomed) from 7 days before the administration of IMP, during the participation in the study and for 7 days prior to any outpatient visit.
* 17. Family history of long QT syndrome or Torsades de Pointes.
* 18. Subjects with poor peripheral venous access.
* 19. Subjects who had a major surgical procedure or significant traumatic injury within 14 days prior to Day -1, or anticipation of the need for major surgery during the study period.
* 20. Subjects with creatinine clearance <60 mL/minute (calculated using Cockcroft-Gault formula) at Screening.
* 21. History of irritable bowel syndrome or other manifestation of abnormal bowel habit (e.g., diarrhoea, constipation).
* 22. Previous exposure to MT-7117 before the administration of IMP in this study.
* 23. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Cmax - maximum observed plasma concentration (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
tmax - time at which Cmax occurs (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
AUC0 t - area under the plasma concentration time curve from time zero to the last measurable concentration (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
AUC0-∞ - area under the plasma concentration-time curve from time zero to infinity (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
t½ - apparent terminal elimination half-life (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
Kel - terminal elimination rate constant (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
CL/F - apparent clearance (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
VZ/F - apparent volume of distribution (plasma and whole blood) | at pre-dose and up to 168 hours post-dose. If collection is extended up to Day 14: at up to 312 hours post-dose.
Total radioactivity in urine and faeces | Day -1 and up to 168 hours post-dose. If collection is extended up to Day 14: up to 312 hours post-dose.
  Ae (urine), Ae (faeces) and Ae (total): amount excreted and cumulative amount excreted in urine, faeces and total (urine and faeces combined).
Total radioactivity in urine and faeces | Day -1 and up to 168 hours post-dose. If collection is extended up to Day 14: up to 312 hours post-dose.
  %Ae (urine), %Ae (faeces) and %Ae (total): amount excreted and cumulative amount excreted in urine, faeces and total (urine and faeces combined) expressed as a percentage of the dose.

SECONDARY OUTCOMES:
Safety and tolerability as measured by incidence of adverse events (AEs) and serious AEs | Up to 14 Days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Mitsubishi Tanabe Pharma Europe Ltd
Locations (1):
- Investigational Centre, United Kingdom, United Kingdom

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Tsuda M, Teng R. Assessment of Potential Drug-Drug Interactions for Novel Oral Melanocortin-1 Receptor Agonist Dersimelagon. Pharmacol Res Perspect. 2025 Feb;13(1):e70069. doi: 10.1002/prp2.70069. PMID 39887900